CLINICAL TRIAL: NCT05887297
Title: Impact of Cognitive Behavioural Therapy for Insomnia on Endocrine Therapy Adherence: a Mixed Methods Pilot Study
Brief Title: Impact of Cognitive Behavioural Therapy for Insomnia on Endocrine Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Responsible Party: Principal Investigator, Sommer Agnew, Principal Investigator, University of Strathclyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UEC23/09
Record Dates: First submitted 2023-05-09; First posted 2023-06-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Breast Cancer; Adherence, Medication; Quality of Life; Survivorship
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms; Medication Adherence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either intervention group or waitlist control. Intervention group will receive CBT-I intervention following randomisation. Waitlist control group will receive CBT-I after all measures have been completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural therapy for insomnia (Experimental): Following randomisation, participants in the intervention group will receive the CBT-I intervention, delivered over 4 weeks.
  Interventions: Behavioral: Cognitive behavioural therapy for insomnia
- Waitlist control (No Intervention): Participants in the waitlist condition will complete all measures at the same timepoints as the intervention group. They will receive the CBT-I intervention after completing the 12-week follow-up assessment. This will then be used as a baseline measure for these participants to compare to their post-intervention and follow-up after receiving the treatment.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy for insomnia — CBT-I is a multi-component, evidence-based intervention which incorporates both cognitive and behavioural techniques to address symptoms of insomnia, aiming to improve satisfaction with the duration and quality of sleep by reducing trouble falling and/or staying asleep. CBT-I will be delivered over 4 weekly 1-hour sessions, via videoconferencing. Session 1 will include psychoeducation about sleep (the relationship between sleep and mental health, the '3P' model of insomnia), and begin to explain components of CBT-I (sleep restriction and relaxation). Session 2 will reinforce previous learning about these components and introduce stimulus control. Session 3 will introduce sleep hygiene and its importance in preventing poor sleep. Session will 4 discuss cognitive therapy techniques and relapse prevention.
  Arms: Cognitive behavioural therapy for insomnia

SUMMARY:
The aim of this study is to investigate the impact of cognitive behavioural therapy for insomnia on adherence to endocrine therapy medication in breast cancer survivors.

DETAILED DESCRIPTION:
Approximately 70% of breast cancer cases are hormone-receptor positive, therefore treatable with endocrine therapy medication. When taken as prescribed, this is effective in reducing the risk of breast cancer recurrence following primary treatment. However, research indicates that nonadherence (not taking medication as prescribed, whether due to forgetfulness or deliberately missing a dose) is an issue, with side effects being a consistent predictor of nonadherence. Sleep problems are one of the most common endocrine therapy side effects. The aim of this study is to explore the influence of cognitive behavioural therapy for insomnia (CBT-I) on endocrine therapy adherence in breast cancer survivors.

Participants will be randomised to 1 of 2 groups: intervention, or waitlist control. Both groups will complete measures of sleep and other endocrine therapy side effects (depression, anxiety, fatigue, musculoskeletal pain, and vasomotor symptoms) at baseline, post-intervention, and 12-week post-randomisation follow-up. Following randomisation, the intervention group will receive 4 weekly group CBT-I sessions remotely through videoconferencing, whereas waitlist control participants will receive the intervention after 12 weeks, once all measures are completed.

Primary outcome will be self-reported endocrine therapy adherence, with secondary outcomes including insomnia symptoms and other endocrine therapy side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Aged 18 or over
* Currently prescribed endocrine therapy medication
* Experience symptoms of insomnia
* Self-reported nonadherent to ET medication (e.g. forgetting to take, or deliberately taking a break from medication)
* Proficient in English language
* Access to videoconferencing

Exclusion Criteria:

* Undertaking shift work (i.e., irregular or night shifts)
* Pregnancy or breastfeeding
* Other unstable physical or mental health problem (including substance misuse)
* Received CBT-I within past 12 months
* Received chemotherapy or radiotherapy within past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Endocrine therapy adherence | 12 weeks
  Primary outcome will be self-reported adherence to endocrine therapy medication, measured using the Medication Adherence Report Scale (MARS-5). Items are scored from 1-5. Responses are summed to create a total ranging from 1-20, with higher scores indicating better adherence.

SECONDARY OUTCOMES:
Insomnia symptoms | 12 weeks
  Severity of insomnia symptoms, measured using the Sleep Condition Indicator. Items are scored from 0-4. Responses are summed to create a total score ranging from 0-32, with higher scores meaning better sleep.
Depressive symptoms | 12 weeks
  Measured using the Patient Health Questionnaire (PHQ-9). Items are scored from 0-3. Responses are summed to create a total score ranging from 0-27, with higher scores meaning more severe depressive symptoms.
Anxiety symptoms | 12 weeks
  Measured using the Generalised Anxiety Disorder Assessment (GAD-7). Items are scored from 0-3. Responses are summed to create a total score ranging from 0-21, with higher scores meaning more severe anxiety.
Fatigue | 12 weeks
  Measured using the Flinders Fatigue Scale (FFS). This measure includes 7 items. Six items are scored from 0-4, whereas item 5 includes a checklist which is scored from 0-7. Responses are summed to create a total score of 0-31.
Musculoskeletal pain | 12 weeks
  Measured using musculoskeletal subscale of Breast Cancer Eight Symptom Scale. This subscale includes 3 items, scored from 1-3. Scores are summed, multiplied by the number of items in the subscale, and then divided by the number of questions answered, with higher scores indicating worse symptoms.
Vasomotor symptoms | 12 weeks
  Measured using vasomotor subscale of Breast Cancer Eight Symptom Scale. This subscale includes 3 items, scored from 1-3. Scores are summed, multiplied by the number of items in the subscale, and then divided by the number of questions answered, with higher scores indicating worse symptoms.
Sleep efficiency | 12 weeks
  The proportion of time spent in bed which is spent sleeping, measured using Consensus sleep diary. This calculated by dividing the time spent sleeping by time spent in bed, then multiplying this by 100 to generate time spent sleeping as a % of time in bed.
Total sleep time | 12 weeks
  Time spent asleep, measured using Consensus sleep diary.
Sleep onset latency | 12 weeks
  Time taken from getting into bed to falling asleep, measured using Consensus sleep diary.
Wake after sleep onset | 12 weeks
  Amount of time spent awake after initially falling asleep, measured using Consensus sleep diary. This is calculated by adding up the length of all night-time awakenings to create a total in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Strathclyde, Glasgow, County (Optional), United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT05887297/Prot_SAP_ICF_000.pdf